CLINICAL TRIAL: NCT06259565
Title: Non-invasive Ventilation and Dexmedetomidine in Critically Ill Adults: An International Pragmatic Randomized Controlled Trial (inDEX Trial)
Brief Title: Non-invasive Ventilation and Dexmedetomidine in Critically Ill Adults
Acronym: inDEX
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Population Health Research Institute (Other)
Responsible Party: Principal Investigator, Kimberley Lewis, Principal Investigator, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4257
Record Dates: First submitted 2023-12-27; First posted 2024-02-14 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Non-Invasive Ventilation
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Patients randomized to the experimental arm will receive dexmedetomidine. We will start the infusion at a mid-range dose of 0.5mcg/kg/h with titration either up or down by 0.1mcg/kg/h every 20-30 minutes to a maximum rate of 1.2mcg/kg/h to maintain light sedation (RASS = -2 to +1 or SAS = 3 to 4). The study drug will always be titrated to the lowest possible dose with preserved effect. Each bag will be composed of two 100 mcg/mL dexmedetomidine vials (2ml vials) mixed in a 96mL 0.9% sodium chloride mini-bag (4mcg/ml) and labeled as per Health Canada guidance for labelling pharmaceutical drugs for use in humans.
  The trial protocol does not allow an initial bolus of dexmedetomidine for safety reasons.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine Intervention (Experimental): Dexmedetomidine (Dex) is an α2-adrenergic agonist sedative commonly used in IMV that promotes patient wakefulness, has no effect on respiratory drive, has important analgesic properties, and reduces delirium.
  Patients randomized to the experimental arm will receive dexmedetomidine. At initiation, a bolus will NOT be administered. In keeping with Health Canada Guidelines, we will start the infusion at a mid-range dose of 0.5mcg/kg/h with titration either up or down by 0.1mcg/kg/h every 20-30 minutes to a maximum rate of 1.2mcg/kg/h to maintain light sedation (RASS = -2 to +1 or SAS 3-4). Each bag will be composed of composed of dexmedetomidine 4mcg/mL(in 0.9% sodium chloride) prepared as a volume of 100mL and labeled as per Health Canada guidance for labelling pharmaceutical drugs for use in humans.
  Interventions: Drug: Dexmedetomidine
- Placebo Control (Placebo Comparator): Those in the control group will receive a placebo that is identical in colour and packaging and at equal volume to the intervention group. Each bag of placebo contains 100mL of 0.9% sodium chloride and labeled as per Health Canada guidance for labelling pharmaceutical drugs for use in humans
  Interventions: Other: Placebo Control

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine (Dex) is an α2-adrenergic agonist sedative commonly used in invasive mechanical ventilation (IMV) that promotes patient wakefulness, has no effect on respiratory drive, has important analgesic properties, and reduces delirium
  Arms: Dexmedetomidine Intervention
Other: Placebo Control — Those in the control group will receive a placebo that is identical in colour and packaging and at equal volume to the intervention group. Each bag of placebo contains 100mL of 0.9% sodium chloride and labeled as per Health Canada guidance for labelling pharmaceutical drugs for use in humans
  Arms: Placebo Control

SUMMARY:
Non-Invasive ventilation (NIV) is a life saving intervention for patients with acute respiratory failure (ARF). Some patients are not able to tolerate the NIV intervention and ultimately fail, requiring the use of invasive mechanical ventilation (IMV) and intubation. Sedation may improve a patient's NIV tolerance. However, this practice has not been adopted by intensivists as the risk of over-sedation resulting in respiratory depression, inability to protect the airway, and inadvertent need for intubation are all large deterrents of sedative use in NIV.

The Non-invasive Ventilation and Dexmedetomidine in Critically Ill Adults: a Pragmatic Randomized Controlled Trial (inDEX) is looking to evaluate the effectiveness of dexmedetomidine compared to placebo in reducing non-invasive ventilation failures in patients admitted to the hospital with acute respiratory failure.

DETAILED DESCRIPTION:
Acute respiratory failure (ARF) is a common reason for admission to an intensive care unit (ICU). Non-invasive positive pressure ventilation (NIV) is a life-saving intervention for selected patients with ARF. Compared to endotracheal intubation and invasive mechanical ventilation (IMV), NIV is safer, less invasive, preferred by most patients, and is associated with a reduced ICU length of stay (LOS), less pneumonia and mortality, and lower healthcare costs.

NIV failure can occur, necessitating IMV. Risk factors associated with NIV failure including intolerance, agitation, and delirium. Sedation is a potential solution for NIV intolerance, however the evidence is sparse and the risk of over-sedation resulting in respiratory depression, inability to protect the airway, and inadvertent need for intubation are all large deterrents.

Dexmedetomidine (Dex) is an α2-adrenergic agonist sedative commonly used in IMV that promotes patient wakefulness, has no effect on respiratory drive, has important analgesic properties, and reduces delirium. The investigators hypothesize that Dex, when compared to placebo, reduces NIV failure in hospitalized adults with ARF and agitation or NIV intolerance.

Overall Goal: To determine if Dex, compared to placebo, reduces the risk of NIV failure in patients that admitted to hospital with acute respiratory failure and are intolerant of NIV.

Target Population: 846 patients will be enrolled into the trial if they meet all the following criteria: 1) ≥18 years old; 2) Receiving any NIV modality for ARF of any etiology; 3) Admitted to ICU, PACU, step-down unit (surgical or medical), or emergency department; 4) Presence of one or more of the following: a) Agitation, b) Patient expresses intolerance or requests removal of NIV secondary to self-reported discomfort, anxiety, or claustrophobia, or c) Other reason that the physician feels the patient is intolerant of NIV or agitated not captured above, or feels that the patient will benefit from sedation (all reasons will be recorded).

Methods: The inDEX trial is a pragmatic, international, multi-centred, stratified, randomized, parallel-group, placebo-controlled trial. Patients, investigators, healthcare team, data collectors, outcome assessors, and the statistician will be blinded to trial arms. The trial will maximize external validity by including patients in a range of hospitals across the world. Patients randomized to the experimental arm will receive Dex while those randomized to the control arm will receive placebo.

Assessment: The primary outcome is NIV failure. The investigators define NIV failure as the proportion that require intubation or have died at 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Patient receiving any NIV modality for acute respiratory failure of any etiology
3. Admitted to ICU, PACU, step-down unit (surgical or medical), or emergency department(with planned admission to a monitored setting) or equivalent unit where hemodynamics and respiratory status can be monitored, and NIV is permitted; and
4. Presence of one or more of the following after optimized NIV treatment:

   1. Agitation (Defined as a Richmond Agitation and Sedation Scale [RASS] score of ≥+2 or a Riker Sedation-Agitation Scale [SAS] score of ≥5) (Appendix 1 Table 2 and Table 3)
   2. Patient expresses intolerance or requests removal of NIV secondary to self-reported discomfort, anxiety, or claustrophobia
   3. Other reason that the physician judges the patient to be intolerant of NIV or agitated, not captured above, or feels that the patient would benefit from titrated sedation for other reasons.

Exclusion Criteria:

1. Absence of a functioning pacemaker with one of the following: a-Persistent bradycardia defined as a heart rate (HR) ≤60bpm; b-Second or third-degree heart block; or c- Tachybrady syndrome
2. Persistent hypotension, defined as a mean arterial pressure (MAP) ≤65mmHg despite volume resuscitation and vasopressors
3. Imminent need for endotracheal intubation as determined by healthcare team
4. Patient's goals of care do not include intubation and IMV
5. Patient is not for vasopressors or inotropic support
6. Death is deemed imminent and inevitable
7. Patient is currently on a dexmedetomidine infusion for a duration of > 12 hours
8. Previously enrolled in the inDEX trial
9. Acute liver failure with hepatic encephalopathy INR > 3 and/or bilirubin > 300
10. Current pregnancy or breast feeding
11. Known allergy to dexmedetomidine
12. Patients receiving Amphotericin B or Diazepam
13. Treating physician does not believe that participation in the trial is in the best interest of the patient (reasons for refusal will be captured)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 846 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
NIV Failure | 28 days
  The primary outcome is NIV failure, defined by either mortality or intubation

SECONDARY OUTCOMES:
Physiologic outcomes: Incidence of delirium | 28 days
  Delirium assessed using the ICU-CAM or ICDSC every 12 hours during NIV and daily thereafter until ICU discharge
Physiologic outcomes: Incidence of agitation | 28 days
  Agitation defined as Richmond Agitation Sedation Scale (RASS) ≥2+ during NIV), where RASS scale ranges from -5 (unrousable) to +4 (combative).
Major morbidity or mortality outcomes: Intubation | 14 days
  Intubation
Major morbidity or mortality outcomes: ICU Mortality | 28 days
  ICU mortality
Major morbidity or mortality outcomes: Hospital Mortality | 90 days
  Hospital Mortality

OTHER OUTCOMES:
Functional Outcome: EQ-5D-5L | 90 days
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  EQ-5D-5L index scores range from -0.59 to 1, where 1 is the best possible health state
Functional Outcome: EQ-VAS | 90 days
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale where the endpoints are labelled 'The best health you can image' and 'The worst health you can image'. The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
  EQ VAS scores range from 0 to 100, where 100 is the best possible health state.
Functional Outcome: Clinical Frailty Scale | 90 days
  The CFS summarizes the overall level of fitness or frailty of an older adult after they had been evaluated by a clinician.
  A score from 1 (very fit) to 9 (terminally ill) is given based on the descriptions and pictographs of activity and functional status.
Hospital outcomes | 90 days
  Hospital Length of Stay (LOS)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberley Lewis, MD, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (6):
- Canada (6):
  - Fraser Health Authority, Surrey, British Columbia
  - Brockville General Hospital, Brockville, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Juravinski Hospital and Cancer Centre, Hamilton, Ontario
  - North York General Hospital, Toronto, Ontario
  - Sinai Health System, Toronto, Ontario